CLINICAL TRIAL: NCT06391242
Title: A Randomized Phase III Trial Comparing Stereotactic Body Radiotherapy to Conventional Palliative Radiotherapy (SBRT) Versus Conventional Palliative Radiotherapy (CRT) for Participants With Painful Non-Spine Bone Metastases
Brief Title: Stereotactic Body Radiotherapy vs Conventional Palliative Radiotherapy for Painful Non-Spine Bone Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC29
Record Dates: First submitted 2024-04-17; First posted 2024-04-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Conventional Radiotherapy (Active Comparator)
  Interventions: Radiation: Standard Conventional Radiotherapy
- Stereotactic Body Radiotherapy (Experimental)
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Standard Conventional Radiotherapy — 20Gy in 5 fractions
  Arms: Standard Conventional Radiotherapy
Radiation: Stereotactic Body Radiotherapy — 30 or 35Gy in 5 fractions
  Arms: Stereotactic Body Radiotherapy

SUMMARY:
This study is being done to answer the following question: Is Stereotactic Body Radiation Therapy or SBRT (a form of radiation therapy which can deliver high doses of radiation to the specific painful area of the body most affected by cancer, while keeping the radiation beams away from the healthy parts of the body that surround the cancer) better for pain relief than the standard treatment of conventional radiation therapy or CRT (a form of radiation therapy which delivers radiation to the painful area but can also negatively affect other parts of the body in the same area)

DETAILED DESCRIPTION:
This is a multi-centre, phase III randomized controlled trial comparing SBRT to conventional palliative EBRT in patients with solid tumours and a dominant painful non-spine bone metastasis as defined by a worst pain score of 2 or greater. 230 participants will be enrolled to the study. Participants will have radiation for 5 treatments (conventional palliative EBRT 20Gy/5; SBRT 30Gy/5 or 35Gy/5) and then will be followed for pain response and radiological progression at 3 and 6 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of solid tumour.
* Patient with a dominant painful non-spine bone metastasis and a worst minimum pain score of 2 using the BPI attributed to that dominant site
* Expected overall survival of greater than 6 months as determined by the treating physician
* Suitable for protocol defined SBRT and CRT.
* Stable pain with no immediate plan to alter analgesic regimen.
* ECOG performance status of 0-2.
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrolment in the trial to document their willingness to participate

Exclusion Criteria:

* Metastases of the hands, feet, cranium or spine (including sacrum) as the dominant/index pain site.
* Bone metastasis arising from a small cell or germ cell.
* Radionuclide therapy within 30 days of randomization.
* Patient treated with prior palliative RT to the dominant painful bone metastasis site (prior radiation exposure is permitted if prior to development of the dominant metastasis and would not influence the applicability of either treatment arm of the current study).
* Received systemic chemotherapy within 1 week of the protocol RT, or who are expected/planned to receive chemotherapy within one week of completing protocol RT.
* Participants with an unstable pathologic fracture at the dominant painful bone metastasis, or for whom surgical fixation would be the preferred intervention if possible.
* Pregnant or lactating individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete pain response utilizing the Cochran-Mantel-Hanzeal test | 27 months

SECONDARY OUTCOMES:
Pain response pattern at 3 months: partial, stable or progressive pain | 27 months
Early (1 month post RT) and late (6 months post RT) CPR and response patterns (partial, stable, and progressive pain); | 27 months
Re-irradiation rate within the 6-month follow-up period | 27 months
Incidence of fracture at the radiation target site | 27 months
Incidence of treatment-related AE rates >/- grade 2 utilizing CTCAE v5 | 27 months
Imaging-based local control rates at 3 and 6 months post-treatment | 27 months
Patient reported outcomes utilizing EORTC QLQ-C30 | 27 months
Patient reported outcomes utilizing EORTC QLQ-BM22 | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Sahgal, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, ON, Canada; Tim Nguyen, Study Chair — London Regional Cancer Program, London, ON, Canada
Locations (7):
- Canada (7):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policies